CLINICAL TRIAL: NCT01815931
Title: Hemolysis in Blood Samples in the ER
Status: Completed | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Olivier T. Rutschmann, MD, MPH, University Hospital, Geneva
Other Study IDs: SU-032013
Record Dates: First submitted 2013-03-19; First posted 2013-03-21 (Estimated); Last update posted 2013-11-11 (Estimated); Status verified 2013-11

CONDITIONS: Hemolysis; Emergency Service, Hospital; Emergencies; Blood Specimen Collection
MeSH Terms: conditions — Hemolysis; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ED patients

SUMMARY:
In this study, we aim to identify risk factors for hemolysis in blood samples drawn in the ED.

ELIGIBILITY:
Inclusion Criteria:

* > 16 years

Exclusion Criteria:

* In vivo hemolysis

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All adult (> 16 y) patients admitted in the emergency departement during the study period
Sampling Method: Non-Probability Sample
Enrollment: 2800 (Actual)
Dates: Start 2013-06; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Hemolysis rate | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Geneva, Geneva, Canton of Geneva, Switzerland